CLINICAL TRIAL: NCT03472924
Title: The Effects of Kinesio Tape® on Arthrogenic Muscle Inhibition and Rate of Torque Development
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient recruitment and enrollment. Reduction in study personnel capacity.
Sponsor: Oregon State University (Other)
Responsible Party: Principal Investigator, Marc Norcross, Associate Professor, Oregon State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7967
Record Dates: First submitted 2018-03-14; First posted 2018-03-21 (Actual); Results first posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-02

CONDITIONS: Neural Inhibition; Injuries, Ankle
Keywords: AMI
MeSH Terms: conditions — Ankle Injuries | interventions — Athletic Tape

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Kinesio Tape (Experimental): Kinesiotaping of the peroneus longus according to the guidelines provided by the Kinesio Taping Association (Kase, K. 2016) followed by standardized set of therapeutic exercises that are commonly implemented in ankle rehabilitation programs.
  Interventions: Device: Kinesiotaping
- Control (No Intervention): Baseline measures followed by standardized set of therapeutic exercises that are commonly implemented in ankle rehabilitation programs, but no use of kinesiotape.

INTERVENTIONS:
Device: Kinesiotaping — The application of Kinesio Tape® (kinesiotaping) according to the guidelines provided by the Kinesio Taping Association (Kase, K. 2016). A 5 cm width strip of Kinesio Tape® (Kinesio TEX Products, NKT-050, Japan) will be applied from origin (the head of the fibula) to insertion (the medial cuneiform and first metatarsal) of the peroneus longus in a longitudinal direction. The proximal anchors will be applied without tension, and the Kinesio Tape® placed on approximately 50% stretch before being applied over the peroneus longus and the distal anchor point.
  Other Names: Kinesio Tape®
  Arms: Kinesio Tape

SUMMARY:
This study evaluates whether the use of Kinesio Tape® in combination with a standard exercise program improves muscle function in individuals with chronic ankle instability. Twenty participants will receive Kinesio Tape® and perform an ankle exercise program, while twenty will perform the ankle exercise program without Kinesio Tape®.

DETAILED DESCRIPTION:
Decreased ability to voluntarily activate the entire motoneuron (MN) pool following joint injury is known as arthrogenic muscle inhibition (AMI), which is commonly quantified by measuring central activation ratio (CAR). AMI is not only observed immediately after joint injury, but has been shown to persist during and after rehabilitation. It is proposed that AMI, by negatively impacting neuromuscular factors such as muscle strength, muscle activation, and rate of torque development (RTD), contributes to a prolonged rehabilitation process and higher risk of re-injury. Unfortunately, AMI cannot be reduced by traditional rehabilitation interventions such as strength training alone. Therefore, it is necessary to identify an intervention that can effectively decrease AMI in order to facilitate improvements in muscle function in individuals with AMI.

Kinesio Tape® is commonly used to facilitate muscle contraction in athletic populations. This elastic therapeutic tape is popular in the athletic setting because it can be applied and used continually during exercise and activities of daily living for up to 2-3 days without restricting movement. It has been suggested that Kinesio Tape® facilitates muscle contraction by inducing increased sensory input via skin stimulation. The tape activates cutaneous mechanoreceptors with the greater afferent feedback thought to improve the efferent output from the central nervous system to the target muscles. While this technique is widely used in the clinical setting to improve muscle function, the facilitative effect of Kinesio Tape® has not been demonstrated- perhaps due to three key limitations of previous investigations. First, previous studies have predominantly recruited healthy participants without muscle function deficits. Therefore, there could have been a ceiling effect whereby there was no observable effect of Kinesio Tape® due to a lack of muscle dysfunction in these healthy individuals. Second, most investigators have generally taken outcome measurements immediately before Kinesio Tape® application and less than 24 hours later. This is much shorter than the 2-3 days that Kinesio Tape® is used clinically and may not be long enough to induce an observable, facilitative effect. Finally, the protocols utilized in previous investigations also failed to mimic clinical practice by not combining Kinesio Tape® application with a therapeutic exercise protocol targeting the inhibited muscle.

Therefore, the purpose of this study is to investigate the effects of prolonged application (> 48hours) of Kinesio Tape® incorporated with a therapeutic exercise protocol on AMI and muscle function. To do so, we will use the peroneus longus muscle in individuals with functional ankle instability (FAI) as a model, given that AMI has been shown to exist in this muscle in individuals with FAI.

The following specific aims will be tested:

Aim#1. To investigate the effect of prolonged application (> 48hours) of Kinesio Tape® incorporated with a therapeutic exercise protocol on AMI of the peroneus longus in individuals with FAI.

Aim#2. To investigate the effect of prolonged application(> 48hours) of Kinesio Tape® incorporated with a therapeutic exercise protocol on peroneus longus muscle function in individuals with FAI.

Our central hypothesis is that prolonged application of Kinesio Tape® in combination with therapeutic exercise will diminish AMI and improve muscle function of the inhibited peroneus longus muscle.

ELIGIBILITY:
Inclusion Criteria:

1. A history of at least one significant ankle sprain on the involved (injured) limb i. The initial sprain must have occurred at least 12 months prior to the study enrollment ii. Was associated with inflammatory symptoms (pain, swelling, etc.) iii. Created at least one interrupted day of desired physical activity.
2. The most recent injury on the involved (injured) ankle must have occurred more than 3 months prior to the study enrollment.
3. A history of the involved (injured) ankle joint 'giving way', and/or recurrent sprain and/or 'feelings of instability' on the involved (injured) limb Participants should report at least 2 episodes of 'giving way' in the 6 months prior to the study enrolment.
4. Be 18-35 years of age
5. Have not had a past allergic reaction to Kinesio Tape®

Exclusion Criteria:

1. Have a history of previous surgeries to the musculoskeletal structures (i.e., bones, joint structures, nerves, etc.) in either lower extremity.
2. Have a history of a fracture in either lower extremity requiring realignment.
3. Had acute injury to the musculoskeletal structures of other joints of either lower extremity in the previous 3 months which impacted joint integrity and function (i.e., sprains, fractures, etc.) and resulted in at least 1 interrupted day of desired physical activity.
4. Are not able to be matched according to our group allocation procedure
5. Have had a past allergic reaction to Kinesio Tape®
6. Currently display symptoms of an acute sprain including swelling, heat, redness, pain, discoloration, and/or loss of range of motion or function
7. Any diagnosed vestibular disorder, Charcot-Marie-Tooth disorder, Ehlers-Danlos, or other hereditary nerve, balance or connective tissue disorder
8. Report a possibility that they may be pregnant as hormonal changes may affect ligamentous laxity
9. Have suffered more than one ankle sprain on the uninvolved limb
10. Have had an ankle sprain on the uninvolved limb within the past 12 months
11. Have episodes of giving way of the ankle on the uninvolved limb besides the single time when they may have sprained this ankle.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc F Norcross, PhD, Principal Investigator — Oregon State University
Locations (1):
- Oregon State University, Corvallis, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akbas E, Atay AO, Yuksel I. The effects of additional kinesio taping over exercise in the treatment of patellofemoral pain syndrome. Acta Orthop Traumatol Turc. 2011;45(5):335-41. doi: 10.3944/AOTT.2011.2403. PMID 22032998
- [Background] Yoshida A, Kahanov L. The effect of kinesio taping on lower trunk range of motions. Res Sports Med. 2007 Apr-Jun;15(2):103-12. doi: 10.1080/15438620701405206. PMID 17578750
- [Background] McVey ED, Palmieri RM, Docherty CL, Zinder SM, Ingersoll CD. Arthrogenic muscle inhibition in the leg muscles of subjects exhibiting functional ankle instability. Foot Ankle Int. 2005 Dec;26(12):1055-61. doi: 10.1177/107110070502601210. PMID 16390639

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Kinesio Tape | Control
Started | 4 | 2
Completed | 3 | 2
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Kinesio Tape | Control | Total
Number analyzed (Participants) | 4 | 2 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 6
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 1 | 0 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in Central Activation Ratio
Description: Ratio between maximal voluntary evertor torque and torque produced following the application of an exogenous electrical stimulus
Time Frame: Change between baseline and 2 days post-intervention
Population: Uneven recruitment and 1 KT participant withdrawn
Measure: Mean (Standard Deviation); unit: Central Activation Torque Ratio
Arm/Group | Kinesio Tape | Control
Number analyzed (Participants) | 3 | 2
Central Activation Torque Ratio | 0.003 (0.024) | 0.015 (0.035)

2. Primary Outcome: Change in Rate of Torque Development
Description: Measure of explosive strength determined by placing a line of best fit to a recorded torque-time curve from onset to 100ms after onset
Time Frame: Change between baseline and 2 days post-intervention
Population: Uneven recruitment and 1 KT participant withdrawn
Measure: Mean (Standard Deviation); unit: Nm/s/kg
Arm/Group | Kinesio Tape | Control
Number analyzed (Participants) | 3 | 2
Nm/s/kg | -0.130 (0.171) | -0.024 (0.010)

3. Secondary Outcome: Change in Maximal Voluntary Isometric Contraction
Description: Measure of maximal voluntary isometric torque that participant can produce
Time Frame: Change between baseline and 2 days post-intervention
Population: Uneven participant recruitment and 1 KT participant withdrawn
Measure: Mean (Standard Deviation); unit: Nm/kg
Arm/Group | Kinesio Tape | Control
Number analyzed (Participants) | 3 | 2
Nm/kg | 0.001 (0.037) | 0.035 (0.043)

ADVERSE EVENTS:
Time Frame: 3 days (Time of kinesotape application to post-testing session 3 days later)
Arm/Group | Kinesio Tape | Control
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/2
Other Adverse Events (participants affected / at risk) | 1/4 | 0/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Kinesio Tape (N=4) | Control (N=2)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Minor skin irritation secondary to Kinseotape

LIMITATIONS AND CAVEATS:
Early termination of the study due inadequate participant enrollment. Results presented are for only 6 total participants and should be intrepreted with extreme caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-07-13): https://cdn.clinicaltrials.gov/large-docs/24/NCT03472924/Prot_001.pdf
  • Informed Consent Form (2017-07-21): https://cdn.clinicaltrials.gov/large-docs/24/NCT03472924/ICF_000.pdf